CLINICAL TRIAL: NCT00814489
Title: A Study to Evaluate GlaxoSmithKline (GSK) Biologicals' Investigational Vaccination Regimen in Healthy Young Adults
Brief Title: Evaluation of Non-typable Haemophilus Influenzae and Pneumococcal Protein Vaccine Formulations in Young Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112076
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2013-07

CONDITIONS: Streptococcus Pneumoniae; Haemophilus Influenzae
Keywords: Non-typable Haemophilus influenzae; protein vaccine; Streptococcus pneumoniae; young adults
MeSH Terms: conditions — Haemophilus Infections | interventions — Engerix-B

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- GSK2254233A Group (Experimental): Subjects received 2 doses of adjuvanted Non-Typable Haemophilus influenza and pneumococcal vaccine GSK2254233A at Months 0 and 2. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK2231395A
- GSK2254232A Group (Experimental): Subjects received 2 doses of non-adjuvanted Non-Typable Haemophilus influenza and pneumococcal vaccine GSK2254232A at Months 0 and 2. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK2231395A
- Engerix Group (Active Comparator): Subjects received 3 doses of Engerix vaccine at Months 0, 2 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: GSK2231395A — Two doses will be administered intramuscularly; one dose at Month 0 and the second dose a Month 2. Two different formulations of this vaccine will be tested.
  Arms: GSK2254232A Group; GSK2254233A Group
Biological: Engerix-B — Two doses will be administered intramuscularly; one dose at Month 0 and the second dose a Month 2.
  Arms: Engerix Group

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of 2 formulations of a non-typable Haemophilus influenzae and pneumococcal candidate vaccine in young adults. Subjects will be vaccinated 2 times in an observer-blind manner with an interval of 2 months. The subjects receiving Engerix-B will receive in an open-manner a third dose of the vaccine at Month 6. The protocol posting has been updated following a protocol amendment.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following amendment of the Protocol, January 2010. The sections impacted are: study design and study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 18 and 40 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Subject without medical history, clinical finding or laboratory finding, which, in the opinion of the investigator, could pose a safety concern or interfere with the protocol.
* If the subject is female, and of childbearing potential, she agrees to use adequate contraception and not become pregnant for the duration of the study.

Exclusion Criteria:

* Pneumonia within 3 years prior to 1st vaccination.
* Invasive Pneumococcal Disease within 3 years prior to 1st vaccination.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period or participation to another pharmaceutical/vaccine study.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccines, with the exception of the influenza vaccine which can be administered >14 days prior to or >14 days following vaccine doses 1 and 2.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* History of reaction or hypersensitivity to any component of the vaccine.
* Any serious, uncontrolled disease likely to interfere with the study as determined by history, physical examination or laboratory screening, as per the judgment of the Investigator.
* Inflammatory processes such as known chronic infections.
* All past or current malignancies and lymphoproliferative disorders.
* Laboratory evidence of haematological and biochemical abnormalities.
* Acute disease at the time of enrolment/vaccination.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Other conditions that the principal investigator judges may interfere with study findings.
* Previous vaccination for hepatitis B. As a portion of the subjects will be randomized to receive Engerix-B comparator, it is important that all subjects meet Engerix-B eligibility criteria.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01-08; Primary Completion 2009-05-04 (Actual); Study Completion 2010-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Karlskrona, Sweden

REFERENCES:
- [Derived] Berglund J, Vink P, Tavares Da Silva F, Lestrate P, Boutriau D. Safety, immunogenicity, and antibody persistence following an investigational Streptococcus pneumoniae and Haemophilus influenzae triple-protein vaccine in a phase 1 randomized controlled study in healthy adults. Clin Vaccine Immunol. 2014 Jan;21(1):56-65. doi: 10.1128/CVI.00430-13. Epub 2013 Oct 30. PMID 24173029

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Started | 15 | 17 | 8
Completed | 13 | 17 | 7
Not Completed | 2 | 0 | 1
Not completed — Other | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK2254233A Group: Subjects received 2 doses of GSK2254233A adjuvanted Non-Typable Haemophilus influenza and pneumococcal vaccine GSK2254233A at Months 0 and 2.The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2254232A Group: Subjects received 2 doses of non-adjuvanted GSK2254232A Non-Typable Haemophilus influenza and pneumococcal vaccine GSK2254232A at Months 0 and 2. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
- Total: Total of all reporting groups
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group | Total
Number analyzed (Participants) | 15 | 17 | 8 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.9 (5.91) | 24.3 (3.69) | 26.6 (5.50) | 25.7 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 5 | 22
  Male | 8 | 7 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local and General Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any solicited local symptom was defined as occurrence of any solicited local symptom regardless of intensity grade.
  Solicited general symptoms assessed were fatigue, gastrointestinal, headache, malaise, myalgia and temperature Any temperature was defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C). For other symptoms: Any = any general symptom reported irrespective of intensity grade and relationship to vaccination.
Time Frame: During a 7-day follow up period after any vaccination
Population: The analysis was based on the Total Vaccinated Cohort, which included all subjects with at least one study vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 15 | 17 | 8
Subjects
  Any pain | 15 | 16 | 4
  Any redness | 10 | 7 | 1
  Any swelling | 6 | 7 | 0
  Any fatigue | 12 | 13 | 5
  Any gastrointestinal | 4 | 6 | 1
  Any headache | 11 | 10 | 5
  Any malaise | 6 | 7 | 2
  Any myalgia | 13 | 8 | 3
  Any temperature | 10 | 7 | 2

2. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AE)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Time Frame: During a 30-day (Days 0-29) follow up period after any vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 15 | 17 | 8
Subjects | 10 | 10 | 6

3. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 to Day 420
Population: The analysis was based on the Total Vaccinated Cohort, which included subjects with at least one study vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 15 | 17 | 8
Subjects | 0 | 0 | 0

4. Primary Outcome: Number of Subjects With Any Biochemical Laboratory Abnormalities
Description: Biochemical parameters assessed in blood samples include alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA) and urea (URE).
  Abnormalities reported include values outside the normal ranges. Time points were presented as before (Pre) or after (Post) Dose 1, 2 or 3.
Time Frame: During a 7-day follow up period after vaccine dose 1 and 2 and at Days 180, 300 and 420
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one study vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 15 | 17 | 8
Subjects
  ALT, Pre Dose 1 (Day 0) [N=2,2,0] | 0 | 0 | NA — This parameter was not measured at Day 0 for subjects in the Engerix Group.
  ALT, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  ALT, Post Dose 1 (Day 60) [N=15,17,7] | 1 | 0 | 0
  ALT, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  ALT, Post Dose 2 (Day 180) [N=14,17,7] | 0 | 1 | 0
  ALT, Post Dose 2 or 3 (Day 300) [N=15,16,6] | 0 | 1 | 0
  ALT, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 2 | 0
  AST, Pre Dose 1 (Day 0) [N=2,3,0] | 0 | 0 | NA — This parameter was not measured at Day 0 for subjects in the Engerix Group.
  AST, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  AST, Post Dose 1 (Day 60) [N=15,17,7] | 1 | 0 | 0
  AST, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  AST, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 2 | 0
  AST, Post Dose 2 or 3 (Day 300) [N=15,16,6] | 0 | 1 | 0
  AST, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  CREA, Pre Dose 1 (Day 0) [N=2,3,0] | 0 | 0 | NA — This parameter was not measured at Day 0 for subjects in the Engerix Group.
  CREA, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  CREA, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  CREA, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  CREA, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  CREA, Post Dose 2 or 3 (Day 300) [N=15,16,5] | 0 | 0 | 0
  CREA, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  URE, Pre Dose 1 (Day 0) [N=2,3,0] | 0 | 0 | NA — This parameter was not measured at Day 0 for subjects in the Engerix Group.
  URE, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  URE, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  URE, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  URE, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  URE, Post Dose 2 or 3 (Day 300) [N=15,16,5] | 0 | 0 | 0
  URE, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Any Hematological Laboratory Abnormalities
Description: Hematological parameters assessed in blood samples include red blood cells (RBC), white blood cells (WBC - including Basophils (BAS), neutrophils (NEU), lymphocytes (LYM), eosinophils (EOS) and monocytes (MON), blood platelets (PLA) and Hemoglobin (HEM). Abnormalities reported include values outside the normal ranges.
  This outcome presents results for RBC, WBC High and Low, PLA and HEM. Time points were presented as before (pre) or after (post) doses 1, 2 or 3.
Time Frame: During a 7-day follow up period after vaccine dose 1 and 2 and at Days 180, 300 and 420.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 15 | 17 | 8
Subjects
  RBC, Pre Dose 1 (Day 0) [N=2,3,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  RBC, Post Dose 1 (Day 7) [N=15,17,8] | 2 | 1 | 1
  RBC, Post Dose 1 (Day 60) [N=15,17,7] | 1 | 4 | 2
  RBC, Post Dose 2 (Day 67) [N=15,17,7] | 3 | 2 | 0
  RBC, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 2 | 0
  RBC, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 1 | 2 | 1
  RBC, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 2 | 1 | 0
  WBC High, Pre Dose 1 (Day 0) [N=2,4,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  WBC High, Post Dose 1 (Day 7) [N=15,17,8] | 1 | 0 | 0
  WBC High, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 1 | 0
  WBC High, Post Dose 2 (Day 67) [N=15,17,7] | 1 | 0 | 0
  WBC High, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 1 | 0
  WBC High, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  WBC High, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  WBC Low, Pre Dose 1 (Day 0) [N=2,4,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  WBC Low, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  WBC Low, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  WBC Low, Post Dose 2 (Day 67) [N=15,17,7] | 1 | 1 | 0
  WBC Low, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  WBC Low, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  WBC Low, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 1 | 0 | 0
  PLA, Pre Dose 1 (Day 0) [N=2,3,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  PLA, Pre Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  PLA, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  PLA, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  PLA, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  PLA, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  PLA, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  HEM, Pre Dose 1 (Day 0) [N=2,3,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  HEM, Post Dose 1 (Day 7) [N=15,17,8] | 1 | 0 | 0
  HEM, Post Dose 1 (Day 60) [N=15,17,7] | 1 | 1 | 1
  HEM, Post Dose 2 (Day 67) [N=15,17,7] | 1 | 0 | 1
  HEM, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 1 | 1
  HEM, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 1 | 0 | 0
  HEM, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Any Hematological Laboratory Abnormalities
Description: Hematological parameters assessed in blood samples include red blood cells (RBC), white blood cells (WBC - including Basophils (BAS), neutrophils (NEU), lymphocytes (LYM), eosinophils (EOS) and monocytes (MON)), blood platelets (PLA) and Hemoglobin (HEM). Abnormalities reported include values outside the normal ranges.
  This outcome presents results for BAS, NEU, LYM, EOS and MON. Time points were presented as before (Pre) or after (Post) Dose 1, 2 or 3.
Time Frame: During a 7-day follow up period after vaccine dose 1 and 2 and at Days 180, 300 and 420.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 15 | 17 | 8
Subjects
  BAS, Pre Dose 1 (Day 0) [N=2,4,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  BAS, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  BAS, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  BAS, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  BAS, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  BAS, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  BAS, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  NEU, Pre Dose 1 (Day 0) [N=2,4,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  NEU, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  NEU, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  NEU, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  NEU, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  NEU, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  NEU, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  LYM, Pre Dose 1 (Day 0) [N=2,4,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  LYM, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  LYM, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  LYM, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  LYM, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  LYM, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  LYM, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  EOS, Pre Dose 1 (Day 0) [N=2,4,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  EOS, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  EOS, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  EOS, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  EOS, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  EOS, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  EOS, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0
  MON, Pre Dose 1 (Day 0) [N=2,4,0] | 0 | 0 | NA — This parameter was not assessed at Day 0 for subjects in the Engerix Group.
  MON, Post Dose 1 (Day 7) [N=15,17,8] | 0 | 0 | 0
  MON, Post Dose 1 (Day 60) [N=15,17,7] | 0 | 0 | 0
  MON, Post Dose 2 (Day 67) [N=15,17,7] | 0 | 0 | 0
  MON, Post Dose 2 (Day 180) [N=15,17,7] | 0 | 0 | 0
  MON, Post Dose 2 or 3 (Day 300) [N=15,16,7] | 0 | 0 | 0
  MON, Post Dose 2 or 3 (Day 420) [N=14,16,7] | 0 | 0 | 0

7. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD), Pneumolysin (Anti-Ply) and Pneumococcal Histidine Triad D (Anti-PhtD)
Description: Concentrations were given as Geometric Mean Concentrations (GMCs). The cut-off values were 112 Luminex Units per milliliter (LU/mL) for Anti-PD, 391 LU/mL for Anti-PhtD and 591 LU/mL for Anti-Ply.
Time Frame: Days 0, 30, 60, 90, 180 and 420.
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who had received at least one dose of study vaccine/comparator and for whom data concerning immunogenicity measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: LU/mL
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 15 | 17 | 7
LU/mL
  Anti-PD, Day 0 [N=15,17,7] | 128.4 [84.3 to 195.5] | 92.3 [63.0 to 135.2] | 286.9 [178.9 to 460.1]
  Anti-PD, Day 30 [N=15,17,7] | 1314.4 [908.5 to 1901.7] | 611.8 [383.2 to 976.5] | 274.9 [173.7 to 435.2]
  Anti-PD, Day 60 [N=15,17,7] | 791.3 [548.4 to 1141.7] | 322.6 [198.3 to 524.8] | 242.9 [149.0 to 395.8]
  Anti-PD, Day 90 [N=15,17,7] | 2142.2 [1224.5 to 3747.6] | 940.9 [534.9 to 1655.0] | 271.2 [173.7 to 423.5]
  Anti-PD, Day 180 [N=14,17,7] | 1351.9 [711.6 to 2568.3] | 416.2 [221.8 to 781.2] | 242.8 [124.8 to 472.5]
  Anti-PD, Day 420 [N=13,16,6] | 943.4 [486.1 to 1830.8] | 278.9 [152.4 to 510.2] | 230.4 [104.8 to 506.9]
  Anti-PhtD, Day 0 [N=15,17,7] | 21128.2 [14752.8 to 30258.6] | 23633.0 [15894.5 to 35139.1] | 18313.4 [10213.3 to 32837.6]
  Anti-PhtD, Day 30 [N=15,17,7] | 78690.3 [52101.6 to 118848.0] | 56628.0 [36231.6 to 88506.4] | 17881.4 [9569.3 to 33413.6]
  Anti-PhtD, Day 60 [N=15,17,7] | 87193.5 [54264.6 to 140104.3] | 58419.9 [36277.8 to 94076.3] | 16396.0 [8813.5 to 30501.9]
  Anti-PhtD, Day 90 [N=15,17,7] | 140774.7 [99455.4 to 199260.3] | 110714.0 [72468.8 to 169142.8] | 20184.0 [10800.8 to 37719.1]
  Anti-PhtD, Day 180 [N=14,17,7] | 87320.6 [61726.8 to 123526.3] | 73013.5 [50712.8 to 105120.8] | 14537.6 [8965.9 to 23571.9]
  Anti-PhtD, Day 420 [N=13,16,7] | 52951.7 [36919.6 to 75945.6] | 52798.1 [36302.4 to 76789.3] | 14432.0 [7243.1 to 28755.7]
  Anti-Ply, Day 0 [N=15,17,7] | 14298.4 [10112.9 to 20216.2] | 14059.5 [9488.5 to 20832.6] | 17523.6 [8747.5 to 35104.6]
  Anti-Ply, Day 30 [N=15,17,7] | 170818.2 [116569.1 to 250313.8] | 106387.7 [50833.5 to 222655.3] | 20190.6 [9177.3 to 44420.5]
  Anti-Ply, Day 60 [N=15,17,7] | 161893.6 [104981.6 to 249658.5] | 87557.0 [41715.7 to 183773.6] | 18387.8 [8281.0 to 40829.5]
  Anti-Ply, Day 90 [N=15,17,7] | 274366.3 [206601.5 to 364357.6] | 163653.4 [92214.9 to 290434.8] | 21144.8 [10650.6 to 41978.8]
  Anti-Ply, Day 180 [N=14,17,7] | 139883.3 [103879.1 to 188366.5] | 91157.5 [53308.3 to 155880.0] | 16737.4 [7740.2 to 36193.1]
  Anti-Ply, Day 420 [N=13,16,7] | 92790.4 [64466.4 to 133558.8] | 59059.5 [34604.5 to 100797.0] | 15832.6 [8103.3 to 30934.3]

8. Secondary Outcome: Mean Number of Influenza-specific Cluster of Differentiation (CD) 4 T-cells.
Description: The mean number was calculated for CD4+ cells stimulated by protein D (PD), pneumococcal histidine triad D (PhtD) or pneumolysin toxoid (dPly), identified as producing T-lymphocyte Helper 1 cells (Th1) versus Th2 cytokines (interferon-gamma (IFN-g) and interleukin-13 (IL-13) respectively, as measured by intracellular staining (ICS) on Peripheral Blood Mononuclear Cells (PBMCs). The outcome presents results for cells producing the following combinations:
  Th1=IFN-g, Th 2=IL13 and/or IL5 and Th17=IL17.
Time Frame: Prior to first vaccination (Day 0), at 14 days post vaccination 1 (Day 14) and 2 (Day 74) and at Day 480.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Groups:
- GSK2254232A Adjuvanted Group: Subjects received 2 doses of adjuvanted Non-Typable Haemophilus influenza and pneumococcal vaccine GSK2254233A at Months 0 and 2. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2254232A Non-adjuvanted Group: Subjects received 2 doses of non-adjuvanted Non-Typable Haemophilus influenza and pneumococcal vaccine GSK2254232A at Months 0 and 2. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
Arm/Group | GSK2254232A Adjuvanted Group | GSK2254232A Non-adjuvanted Group | Engerix Group
Number analyzed (Participants) | 14 | 17 | 7
T-cells/million cells
  Th 1, PD specific, Day 0 [N=14,17,7] | 13.4 (32.1) | 6.8 (23.5) | 10.4 (21.4)
  Th 1, PD specific, Day 14 [N=13,17,6] | 22.2 (42.5) | 7.7 (35.9) | 7.2 (29.0)
  Th 1, PD specific, Day 74 [N=13,17,7] | 157.6 (239.1) | 37.9 (39.9) | -6.0 (32.1)
  Th 1, PD specific, Day 480 [N=11,17,6] | 8.0 (38.5) | -5.8 (23.0) | 58.7 (94.4)
  Th 1, PhtD specific, Day 0 [N=14,17,7] | 0.0 (30.8) | -2.4 (21.4) | -5.1 (16.6)
  Th 1, PhtD specific, Day 14 [N=13,17,6] | 177.5 (263.9) | 61.6 (122.3) | 6.3 (20.1)
  Th 1, PhtD specific, Day 74 [N=13,17,7] | 552.3 (374.0) | 305.4 (294.4) | -1.9 (34.9)
  Th 1, PhtD specific, Day 480 [N=11,17,6] | 34.0 (65.1) | 16.8 (37.4) | 14.5 (25.9)
  Th 1, dPly specific, Day 0 [N=14,17,7] | 75.9 (63.1) | 27.0 (52.6) | 133.4 (209.9)
  Th 1, dPly specific, Day 14 [N=13,17,6] | 233.1 (199.0) | 99.3 (163.7) | 92.5 (138.8)
  Th 1, dPly specific, Day 74 [N=13,17,7] | 576.1 (348.2) | 214.8 (235.5) | 76.7 (90.6)
  Th 1, dPly specific, Day 480 [N=11,17,6] | 14.9 (33.8) | 0.8 (22.1) | 8.5 (13.4)
  Th 2, PD specific, Day 0 [N=14,17,7] | 24.6 (287.7) | -35.4 (328.2) | 267.3 (887.7)
  Th 2, PD specific, Day 14 [N=13,17,6] | -46.1 (350.3) | 40.0 (120.7) | 381.5 (1016.8)
  Th 2, PD specific, Day 74 [N=13,17,7] | -56.1 (183.0) | -42.0 (265.8) | -43.6 (242.6)
  Th 2, PD specific, Day 480 [N=11,17,6] | 1.1 (141.7) | 13.2 (176.1) | 161.0 (394.8)
  Th 2, PhtD specific, Day 0 [N=14,17,7] | -82.4 (212.4) | -15.6 (305.5) | 238.1 (1001.4)
  Th 2, PhtD specific, Day 14 [N=13,17,6] | -72.7 (373.4) | -47.0 (242.2) | 339.8 (1056.8)
  Th 2, PhtD specific, Day 74 [N=13,17,7] | -100.8 (245.0) | -100.9 (252.9) | -125.6 (453.7)
  Th 2, PhtD specific, Day 480 [N=11,17,6] | 14.9 (139.4) | -8.9 (103.0) | 196.2 (351.7)
  Th 2, dPly specific, Day 0 [N=14,17,7] | -76.3 (212.4) | -31.2 (236.8) | 256.0 (1009.3)
  Th 2, dPly specific, Day 14 [N=13,17,6] | -2.4 (236.8) | -11.5 (128.3) | 407.2 (1227.7)
  Th 2, dPly specific, Day 74 [N=13,17,7] | -4.9 (335.7) | -15.7 (150.3) | -126.9 (271.5)
  Th 2, dPly specific, Day 480 [N=11,17,6] | 6.9 (183.4) | -14.7 (146.5) | 195.0 (414.8)
  Th 17, PD specific, Day 0 [N=12,17,7] | 24.7 (80.1) | 17.5 (39.7) | 8.0 (23.0)
  Th 17, PD specific, Day 14 [N=12,17,6] | 19.5 (58.6) | -4.8 (42.7) | -5.5 (71.0)
  Th 17, PD specific, Day 74 [N=12,17,7] | 31.1 (65.2) | 16.2 (66.7) | -17.0 (52.8)
  Th 17, PD specific, Day 480 [N=11,17,6] | 13.5 (34.1) | -4.6 (18.7) | 7.3 (15.3)
  Th 17, PhtD specific, Day 0 [N=12,17,7] | 23.4 (76.5) | 29.5 (56.4) | 12.4 (41.5)
  Th 17, PhtD specific, Day 14 [N=12,17,6] | 70.5 (94.3) | 26.1 (52.9) | 2.4 (49.9)
  Th 17, PhtD specific, Day 74 [N=12,17,7] | 360.8 (267.3) | 114.1 (112.3) | -10.1 (45.3)
  Th 17, PhtD specific, Day 480 [N=11,17,6] | 7.6 (44.9) | -0.5 (28.1) | 9.8 (20.2)
  Th 17, dPly specific, Day 0 [N=12,17,7] | 80.3 (83.0) | 63.9 (79.4) | 122.1 (158.8)
  Th 17, dPly specific, Day 14 [N=12,17,6] | 141.1 (90.5) | 95.4 (88.9) | 88.7 (57.5)
  Th 17, dPly specific, Day 74 [N=12,17,7] | 256.3 (137.3) | 169.9 (125.6) | 82.3 (83.0)
  Th 17, dPly specific, Day 480 [N=11,17,6] | 6.9 (30.7) | 14.0 (26.4) | 10.2 (19.3)

9. Secondary Outcome: Mean Number of Influenza-specific Cluster of Differentiation (CD) 8 T-cells.
Description: The mean number was calculated for CD8+ cells stimulated by protein D (PD), pneumococcal histidine triad D (PhtD) and pneumolysin toxoid (dPly) and expressing the following citokine combinations:
  C1= at least interleukin 2 (IL2), tumor necrosis factor alpha (TNFa) and/or interferon-gamma (IFNg) and C2= at least interleukin 17 (IL17).
Time Frame: Prior to first vaccination (Day 0), at 14 days post vaccination 1 (Day 14) and 2 (Day 74) and at Day 480.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Number analyzed (Participants) | 14 | 17 | 7
T-cells/million cells
  C1, PD specific, Day 0 [N=14,17,7] | -65.0 (166.5) | 28.0 (115.3) | 3.3 (218.3)
  C1, PD specific, Day 14 [N=13,17,6] | -164.8 (247.9) | -20.7 (109.2) | -44.3 (224.5)
  C1, PD specific, Day 74 [N=13,17,7] | -133.3 (225.1) | 7.9 (238.8) | -67.1 (162.7)
  C1, PD specific, Day 480 [N=11,17,6] | -9.5 (525.9) | 68.1 (373.3) | 32.7 (77.3)
  C1, PhtD specific, Day 0 [N=14,17,7] | 36.8 (276.2) | 53.5 (154.8) | 68.6 (271.0)
  C1, PhtD specific, Day 14 [N=13,17,6] | -53.2 (277.0) | 52.9 (170.8) | -54.3 (190.7)
  C1, PhtD specific, Day 74 [N=13,17,7] | -41.2 (269.3) | 122.5 (244.6) | -7.4 (229.8)
  C1, PhtD specific, Day 480 [N=11,17,6] | 4.6 (517.1) | 105.6 (216.7) | 84.7 (114.5)
  C1, dPly specific, Day 0 [N=14,17,7] | -25.2 (188.5) | 15.3 (129.5) | -14.0 (192.1)
  C1, dPly specific, Day 14 [N=13,17,6] | 5.0 (267.1) | -29.8 (208.2) | -104.0 (220.2)
  C1, dPly specific, Day 74 [N=13,17,7] | -29.8 (253.7) | 41.6 (226.5) | -88.1 (182.3)
  C1, dPly specific, Day 480 [N=11,17,6] | -219.1 (655.0) | 58.1 (230.8) | -15.2 (114.2)
  C2, PD specific, Day 0 [N=12,17,7] | -19.0 (150.8) | 74.5 (195.7) | 38.7 (79.5)
  C2, PD specific, Day 14 [N=12,17,6] | 81.8 (105.4) | 8.2 (98.8) | -35.2 (77.5)
  C2, PD specific, Day 74 [N=12,17,7] | 19.0 (69.5) | -11.9 (149.0) | 21.9 (81.1)
  C2, PD specific, Day 480 [N=11,17,6] | -18.9 (91.9) | 103.5 (236.9) | 78.0 (110.9)
  C2, PhtD specific, Day 0 [N=12,17,7] | -30.4 (144.8) | 56.0 (160.6) | 64.7 (106.9)
  C2, PhtD specific, Day 14 [N=12,17,6] | 28.8 (121.9) | 58.8 (130.8) | 15.7 (146.4)
  C2, PhtD specific, Day 74 [N=12,17,7] | 134.3 (321.7) | 20.5 (118.6) | 11.3 (68.2)
  C2, PhtD specific, Day 480 [N=11,17,6] | 7.9 (60.0) | 37.8 (233.5) | 109.8 (210.1)
  C2, dPly specific, Day 0 [N=12,17,7] | -45.8 (119.5) | 31.0 (110.0) | 15.6 (83.3)
  C2, dPly specific, Day 14 [N=12,17,6] | -4.6 (54.0) | 66.2 (124.1) | 1.9 (145.1)
  C2, dPly specific, Day 74 [N=12,17,7] | 7.3 (74.0) | -30.5 (82.2) | -17.1 (62.5)
  C2, dPly specific, Day 480 [N=11,17,6] | -3.7 (150.5) | 38.7 (174.5) | 50.3 (66.1)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected up to Day 420, unsolicited adverse events during a 30-day period after each vaccine dose and solicited symptoms during a 7-day period after each vaccine dose.
Arm/Group | GSK2254233A Group | GSK2254232A Group | Engerix Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/8
Other Adverse Events (participants affected / at risk) | 15/15 | 17/17 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2254233A Group (N=15) | GSK2254232A Group (N=17) | Engerix Group (N=8)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chills (General disorders) | 4 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Injection site reaction (General disorders) | 2 | 2 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Tonsilitis (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain (General disorders) | 15 | 16 | 4
Redness (General disorders) | 10 | 7 | 1
Swelling (General disorders) | 6 | 7 | 0
Fatigue (General disorders) | 12 | 13 | 5
Gastrointestinal symptoms (General disorders) | 4 | 6 | 1
Headache (General disorders) | 11 | 10 | 5
Malaise (General disorders) | 6 | 7 | 2
Myalgia (General disorders) | 13 | 8 | 3
Fever (General disorders) | 10 | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.